CLINICAL TRIAL: NCT06666790
Title: DermaSensor Postmarket Surveillance Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DermaSensor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Screening
Other Study IDs: CSP-24-0002
Record Dates: First submitted 2024-10-28; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Melanoma, Skin
Keywords: medical device; skin cancer detection; elastic scattering spectroscopy
MeSH Terms: conditions — Melanoma | interventions — Radionuclide Imaging

STUDY DESIGN:
Intervention Model Description: Enrolled lesions are assessed without and then with the device result as basis for study investigator decision to biopsy or monitor a potentially malignant lesion.
Who Masked: Investigator
Masking Description: Investigator unaided (i.e., blinded/masked) assessment followed by aided assessment of each lesion's malignancy risk.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Clinical assessment only (No Intervention): Lesions assessed as clinically suspicious by primary care investigator who make diagnostic and management decision to biopsy without ESS device output
- Clinical assessment with device output (Experimental): Lesions assessed as clinically suspicious by primary care investigator who make diagnostic and management decision to biopsy with ESS device output
  Interventions: Device: Scan with elastic scattering spectroscopy device to assess risk of malignancy

INTERVENTIONS:
Device: Scan with elastic scattering spectroscopy device to assess risk of malignancy — Elastic scattering spectroscopy device uses a spectrum of light reflectance to compare suspicious lesion signature to that of previously scanned lesions with known benign or malignant pathology
  Arms: Clinical assessment with device output

SUMMARY:
The objective of this study is to evaluate the sensitivity of the DermaSensor device and Investigators when used on skin lesions concerning for melanoma.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women of any ethnic group aged 40 and older
2. Primary skin lesion suspicious for melanoma
3. Patient is willing and able to read, understand, and sign the informed consent form (ICF)

Exclusion Criteria:

1. Lesion is not accessible to the DermaSensor device Handheld Unit and tip (e.g., inside ears, under nails, etc.)
2. Lesion is on areas of psoriasis, eczema, acne, or similar inflammatory skin conditions that may impede appropriate DermaSensor device tip placement on the lesion.
3. Lesion is greater than 15mm in diameter at the widest point.
4. Lesion has a targeted area less than 2.5mm in diameter where the DermaSensor device tip cannot be placed entirely within the border of the targeted area of the lesion.
5. Lesion has no contiguous area of at least 2.5mm due to ulceration, erosion or liquid discharge (e.g., blood).
6. Lesion is covered by a crust or scale, and lesion surface cannot be cleared of crust or scale such that there is a contiguous area of at least 2.5mm of cleared intact skin that is free of any crust, ulceration, erosion or liquid discharge (e.g., blood).
7. Lesion is obstructed by foreign matter that cannot be non-invasively removed (e.g., tattoo, splinter, etc.)
8. Lesion is not completely cleared of (i.e., free of any remaining residue) dermoscopy oils, makeup, sunscreen, other topical solutions or powders, markings, and staining treatments (e.g., iodine).
9. Lesion is located on acral skin (e.g., sole or palms).
10. Lesion is located within 10mm of the eye.
11. Lesion is on or adjacent to scars, areas previously biopsied, or areas subjected to any past surgical intervention.
12. Lesion is located on mucosal surfaces (e.g. genitals, lips).
13. Lesion is located in an area with acute sunburn.
14. Dementia or other neurologic, physical or psychological limitation that would prevent the patient from signing informed consent and/or completing any required follow-up visits

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2027-04-11 (Estimated); Study Completion 2027-09-10 (Estimated)

PRIMARY OUTCOMES:
Device Sensitivity | 39 months

CONTACTS AND LOCATIONS:
Overall Officials: Gary Slatko, MD, MBA, Study Chair — DermaSensor, Inc.
Locations (2):
- United States (2):
  - Velocity, New Smyrna Beach, Florida
  - West Clinical Research, Morehead City, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided